CLINICAL TRIAL: NCT00003389
Title: A Randomized Phase III Trial of ABVD Versus Stanford V (+/-) Radiation Therapy in Locally Extensive and Advanced Stage Hodgkin's Disease
Brief Title: Combination Chemotherapy With or Without Radiation Therapy in Treating Patients With Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066386; E2496 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine; Vincristine; Mechlorethamine; Etoposide; Podophyllotoxin; Prednisone; Cyclophosphamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (ABVD) (Experimental): Arm A (ABVD): Patients receive doxorubicin (25 mg/m²), bleomycin (10 u/m²), vinblastine (6 mg/m²), and dacarbazine (375 mg/m²) intravenously (IV) on days 1 and 15. Courses repeat every 28 days. Patients are restaged after 4 courses. Patients who are in complete remission receive 2 additional courses. Patients with a partial response or less are evaluated after 6 courses, and if there is an ongoing response, patients may receive 2 additional courses for a total of 8. If no ongoing response is observed, patients are removed from the study. All patients with massive mediastinal disease, regardless of stage, receive radiotherapy 2-3 weeks after completion of chemotherapy.
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Drug: Dacarbazine; Radiation: Radiotherapy
- Arm B (Stanford V) (Active Comparator): Arm B (Stanford V): Patients receive Stanford V chemotherapy comprising doxorubicin (25 mg/m²) and vinblastine (6 mg/m²) IV on day 1 of weeks 1, 3, 5, 7, 9, and 11; vincristine (1.4 mg/m²) and bleomycin (5 u/m²) IV on day 1 of weeks 2, 4, 6, 8, 10, and 12; mechlorethamine (6 mg/m²) IV on day 1 of weeks 1, 5, and 9 (if mechlorethamine is unavailable, may substitute with cyclophosphamide [375 mg/m²] IV); etoposide (60 mg/m²) IV on days 1 and 2 of weeks 3, 7, and 11; and oral prednisone (40 mg/m²) every other day of weeks 1-9 followed by a taper. All patients with bulky disease receive radiotherapy 2-3 weeks after completion of chemotherapy.
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Drug: Vincristine; Drug: Mechlorethamine; Drug: Etoposide; Drug: Prednisone; Drug: Cyclophosphamide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Doxorubicin — given IV
  Other Names: Adriamycin; Rubex; Adriamycin RDF; Adriamycin PFS; hydroxydaunorubicin; hydroxydaunomycin; ADR
Drug: Bleomycin — given IV
  Other Names: Blenoxane; BLM; Bleo
Drug: Vinblastine — given IV
  Other Names: Velban; vinblastine sulfate; vincaleukoblastine; VLB; Velsar; Alkaban AQ
Drug: Dacarbazine — given IV
  Other Names: DTIC; DTIC-Dome; DIC; imidazole carboxamide; dimethyl triazeno imidazole carboxamide
  Arms: Arm A (ABVD)
Drug: Vincristine — given IV
  Other Names: Oncovin; Vincasar PFS; vincristine sulfate; VCR; leurocristine; LCR
  Arms: Arm B (Stanford V)
Drug: Mechlorethamine — given IV
  Other Names: Mustargen; nitrogen mustard
  Arms: Arm B (Stanford V)
Drug: Etoposide — given IV
  Other Names: VP-16; VePesid; VP-16-213; EPEG; epipodophyllotoxin
  Arms: Arm B (Stanford V)
Drug: Prednisone — taken orally
  Other Names: Deltasone; Orasone; Medicorten; Panasol-S; Liquid-Pred
  Arms: Arm B (Stanford V)
Drug: Cyclophosphamide — given IV
  Other Names: Cytoxan; Neosar; CTX; CPM
  Arms: Arm B (Stanford V)
Radiation: Radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining more than one drug with radiation therapy may kill more cancer cells. It is not yet known which combination chemotherapy regimen is most effective in treating Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying two different combination chemotherapy regimens and comparing how well they work, with or without radiation therapy, in treating patients with Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the failure-free survival of patients with locally extensive or advanced Hodgkin's lymphoma treated with doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) vs doxorubicin, vinblastine, vincristine, bleomycin, mechlorethamine, etoposide, and prednisone (Stanford V) with or without radiotherapy.
* Compare the overall survival and freedom from progression in these patients at 5 and 10 years after treatment with these regimens.
* Compare pulmonary function, incidence of second cancers, reproductive function, and deaths from causes other than Hodgkin's lymphoma in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to number of adverse risk factors (0-2 vs 3-7), disease characteristics (locally extensive vs advanced) and time of entry (before addendum 6 vs. after addendum 6). Patients are randomized to 1 of 2 treatment arms.

* Arm A (ABVD): Patients receive doxorubicin (25 mg/m²), bleomycin (10 u/m²), vinblastine (6 mg/m²), and dacarbazine (375 mg/m²) IV on days 1 and 15. Courses repeat every 28 days. Patients are restaged after 4 courses. Patients who are in complete remission receive 2 additional courses. Patients with a partial response or less are evaluated after 6 courses, and if there is an ongoing response, patients may receive 2 additional courses for a total of 8. If no ongoing response is observed, patients are removed from the study. All patients with massive mediastinal disease, regardless of stage, receive radiotherapy 2-3 weeks after completion of chemotherapy.
* Arm B (Stanford V): Patients receive Stanford V chemotherapy comprising doxorubicin (25 mg/m²) and vinblastine (6 mg/m²) IV on day 1 of weeks 1, 3, 5, 7, 9, and 11; vincristine (1.4 mg/m²) and bleomycin (5 u/m²) IV on day 1 of weeks 2, 4, 6, 8, 10, and 12; mechlorethamine (6 mg/m²) IV on day 1 of weeks 1, 5, and 9 (if mechlorethamine is unavailable, may substitute with cyclophosphamide [375 mg/m²] IV); etoposide (60 mg/m²) IV on days 1 and 2 of weeks 3, 7, and 11; and oral prednisone (40 mg/m²) every other day of weeks 1-9 followed by a taper. All patients with bulky disease receive radiotherapy 2-3 weeks after completion of chemotherapy.

Patients are followed every 2 months for 1 year, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 850 patients will be accrued for this study within 4.3 years.

ELIGIBILITY:
Inclusion criteria:

* Histologically proven previously untreated classical Hodgkin's lymphoma
* The following stages are eligible:

  * Locally extensive: Stage I-IIA/B with massive mediastinal adenopathy
  * Advanced: Stage III or IV
* Measurable or evaluable disease
* Age of 16 and over
* ECOG Performance status 0-2
* Disease-free of prior invasive malignancies for >5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* White blood cell (WBC) at least 4,000/mm³, (unless documented bone marrow involvement)
* Platelet count at least 100,000/mm³ (unless documented bone marrow involvement)
* Bilirubin no greater than 5.0 mg/dL
* Creatinine no greater than 2.0 mg/dL
* Ejection fraction determination recommended if over age 50 and/or have a history of cardiac disease
* Fertile patients must use effective contraception
* Prior corticosteroids allowed
* Prior surgery allowed

Exclusion criteria:

* Pregnant or nursing
* Prior radiotherapy
* Prior chemotherapy
* Human immunodeficiency virus (HIV) positive

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 1999-06-17 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Horning, MD, Study Chair — Stanford University
Locations (539):
- United States (517):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Eden Medical Center, Castro Valley, California
  - Mount Diablo Regional Cancer Center, Concord, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Saint Rose Hospital, Hayward, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Memorial Medical Center Cancer Services, Modesto, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - M.D. Anderson Cancer Center - Orlando, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Northwest Medical Specialist, PC, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Medical Consultants, P. C. at Ball Cancer Center, Muncie, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, P. C., Ames, Iowa
  - Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Franklin Medical Center, Greenfield, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Frisbie Memorial Hospital, Rochester, New Hampshire
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Mountainside Hospital Cancer Center, Montclair, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oswego Hospital, Oswego, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Jewish Hospital Cancer Center, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Comanche County Memorial Hospital, Lawton, Oklahoma
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates, Scranton, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Baptist Regional Cancer Center at Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Mount Ascutney Hospital, Windsor, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Washington Hematology-Oncology Specialists, Yakima, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Medical Center - Fish Hatchery, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (21):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - St. Catharines General Hospital at Niagara Health System, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Gordon LI, Hong F, Fisher RI, Bartlett NL, Connors JM, Gascoyne RD, Wagner H, Stiff PJ, Cheson BD, Gospodarowicz M, Advani R, Kahl BS, Friedberg JW, Blum KA, Habermann TM, Tuscano JM, Hoppe RT, Horning SJ. Randomized phase III trial of ABVD versus Stanford V with or without radiation therapy in locally extensive and advanced-stage Hodgkin lymphoma: an intergroup study coordinated by the Eastern Cooperative Oncology Group (E2496). J Clin Oncol. 2013 Feb 20;31(6):684-91. doi: 10.1200/JCO.2012.43.4803. Epub 2012 Nov 26. PMID 23182987
- [Derived] Advani RH, Hong F, Fisher RI, Bartlett NL, Robinson KS, Gascoyne RD, Wagner H Jr, Stiff PJ, Cheson BD, Stewart DA, Gordon LI, Kahl BS, Friedberg JW, Blum KA, Habermann TM, Tuscano JM, Hoppe RT, Horning SJ. Randomized Phase III Trial Comparing ABVD Plus Radiotherapy With the Stanford V Regimen in Patients With Stages I or II Locally Extensive, Bulky Mediastinal Hodgkin Lymphoma: A Subset Analysis of the North American Intergroup E2496 Trial. J Clin Oncol. 2015 Jun 10;33(17):1936-42. doi: 10.1200/JCO.2014.57.8138. Epub 2015 Apr 20. PMID 25897153
- [Derived] Kanakry JA, Li H, Gellert LL, Lemas MV, Hsieh WS, Hong F, Tan KL, Gascoyne RD, Gordon LI, Fisher RI, Bartlett NL, Stiff P, Cheson BD, Advani R, Miller TP, Kahl BS, Horning SJ, Ambinder RF. Plasma Epstein-Barr virus DNA predicts outcome in advanced Hodgkin lymphoma: correlative analysis from a large North American cooperative group trial. Blood. 2013 May 2;121(18):3547-53. doi: 10.1182/blood-2012-09-454694. Epub 2013 Feb 5. PMID 23386127
- [Derived] Evens AM, Hong F, Gordon LI, Fisher RI, Bartlett NL, Connors JM, Gascoyne RD, Wagner H, Gospodarowicz M, Cheson BD, Stiff PJ, Advani R, Miller TP, Hoppe RT, Kahl BS, Horning SJ. The efficacy and tolerability of adriamycin, bleomycin, vinblastine, dacarbazine and Stanford V in older Hodgkin lymphoma patients: a comprehensive analysis from the North American intergroup trial E2496. Br J Haematol. 2013 Apr;161(1):76-86. doi: 10.1111/bjh.12222. Epub 2013 Jan 29. PMID 23356491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 22, 1999 and June 15, 2006, 854 participants were enrolled. The first patient accrued was on June 17, 1999.
Groups:
- Arm A (ABVD): Arm A (ABVD): Patients receive doxorubicin (25 mg/m²), bleomycin (10 u/m²), vinblastine (6 mg/m²), and dacarbazine (375 mg/m²) intravenously (IV) on days 1 and 15. Courses repeat every 28 days. Patients are restaged after 4 courses. Patients who are in complete remission receive 2 additional courses. Patients with a partial response or less are evaluated after 6 courses, and if there is an ongoing response, patients may receive 2 additional courses for a total of 8. If no ongoing response is observed, patients are removed from the study. All patients with massive mediastinal disease, regardless of stage, receive radiotherapy 2-3 weeks after completion of chemotherapy.
  Doxorubicin: given IV
  Bleomycin: given IV
  Vinblastine: given IV
  Dacarbazine: given IV
  Radiotherapy
- Arm B (Stanford V): Arm B (Stanford V): Patients receive Stanford V chemotherapy comprising doxorubicin (25 mg/m²) and vinblastine (6 mg/m²) IV on day 1 of weeks 1, 3, 5, 7, 9, and 11; vincristine (1.4 mg/m²) and bleomycin (5 u/m²) IV on day 1 of weeks 2, 4, 6, 8, 10, and 12; mechlorethamine (6 mg/m²) IV on day 1 of weeks 1, 5, and 9 (if mechlorethamine is unavailable, may substitute with cyclophosphamide [375 mg/m²] IV); etoposide (60 mg/m²) IV on days 1 and 2 of weeks 3, 7, and 11; and oral prednisone (40 mg/m²) every other day of weeks 1-9 followed by a taper. All patients with bulky disease receive radiotherapy 2-3 weeks after completion of chemotherapy.
  Doxorubicin: given IV
  Bleomycin: given IV
  Vinblastine: given IV
  Vincristine: given IV
  Mechlorethamine: given IV
  Etoposide: given IV
  Prednisone: taken orally
  Cyclophosphamide: given IV
  Radiotherapy
Period: Overall Study
Arm/Group | Arm A (ABVD) | Arm B (Stanford V)
Started | 428 | 426
Treated Pts w/ Toxicity Data Available | 414 | 422
Eligible Patients | 395 | 399
Completed | 330 | 366
Not Completed | 98 | 60
Not completed — Disease progression | 6 | 1
Not completed — Adverse Event | 13 | 2
Not completed — Death | 0 | 3
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Alternative therapy | 2 | 1
Not completed — Complicating disease | 1 | 0
Not completed — Off-treatment reason missing | 31 | 21
Not completed — Ineligible | 33 | 27

BASELINE CHARACTERISTICS:
Population: Eligible patients are included in the primary analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (ABVD) | Arm B (Stanford V) | Total
Number analyzed (Participants) | 395 | 399 | 794
Age, Continuous [Median (Full Range); unit: years] | 33 [18 to 83] | 33 [16 to 83] | 33 [16 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 182 | 369
  Male | 208 | 217 | 425
Region of Enrollment [Number; unit: participants]
  Canada | 46 | 50 | 96
  United States | 349 | 349 | 698

OUTCOME MEASURES:

1. Primary Outcome: Failure-free Survival at 5 Years
Description: Failure-free survival is defined as the time from randomization to the earlier of progression/relapse or death. The 5-year failure-free survival is the probability a patient is failure-free and survives 5 years.
  Progression is defined as an increase in size of 25% of the sum of the products of the pretreatment measurements or appearance of new lesions. Significant enlargement of the liver or spleen is evidence of progression. A significant increase in size is defined as > 2.0 cm in distance between costal margin and the inferior margin of either organ.
  Relapse is defined as the re-appearance of any clinical evidence of Hodgkin's disease in a patient who has had a complete response. Relapse for partial responders is defined as progressive disease relative to disease status during the partial remission.
Time Frame: Assessed every 2 months if patient is < 1 year from study entry, every 3 months for the second year, every 4 months for the third year, every 6 months for years 4 and 5
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (ABVD) | Arm B (Stanford V)
Number analyzed (Participants) | 395 | 399
Proportion of patients | 0.74 [0.69 to 0.79] | 0.71 [0.66 to 0.76]
Statistical Analysis 1: Comparison: Arm A (ABVD) vs Arm B (Stanford V); Test type: Superiority or Other; p = 0.32, Log Rank; Stratified log rank test was performed

2. Secondary Outcome: 5-year Overall Survival
Description: Overall survival is defined as the time from randomization to death or last known alive. The 5-year survival rate is the probability a patient survives 5 years.
Time Frame: Assessed every 2 months if patient is < 1 year from study entry, every 3 months for the second year, every 4 months for the third year, every 6 months for years 4 and 5, and yearly for 5 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (ABVD) | Arm B (Stanford V)
Number analyzed (Participants) | 395 | 399
Proportion of patients | 0.88 [0.85 to 0.92] | 0.88 [0.84 to 0.91]
Statistical Analysis 1: Comparison: Arm A (ABVD) vs Arm B (Stanford V); Test type: Superiority or Other; p = 0.86, Log Rank; Stratified log rank test was performed

3. Secondary Outcome: Incidence of Second Cancers
Description: Number of patients who developed second primary cancers
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Arm A (ABVD) | Arm B (Stanford V)
Number analyzed (Participants) | 395 | 399
participants | 15 | 19

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment.
Groups:
- Arm A (ABVD): Patients receive doxorubicin (25 mg/m²), bleomycin (10 u/m²), vinblastine (6 mg/m²), and dacarbazine (375 mg/m²) intravenously (IV) on days 1 and 15. Courses repeat every 28 days. Patients are restaged after 4 courses. Patients who are in complete remission receive 2 additional courses. Patients with a partial response or less are evaluated after 6 courses, and if there is an ongoing response, patients may receive 2 additional courses for a total of 8. If no ongoing response is observed, patients are removed from the study. All patients with massive mediastinal disease, regardless of stage, receive radiotherapy 2-3 weeks after completion of chemotherapy.
- Arm B (Stanford V): Patients receive Stanford V chemotherapy comprising doxorubicin (25 mg/m²) and vinblastine (6 mg/m²) IV on day 1 of weeks 1, 3, 5, 7, 9, and 11; vincristine (1.4 mg/m²) and bleomycin (5 u/m²) IV on day 1 of weeks 2, 4, 6, 8, 10, and 12; mechlorethamine (6 mg/m²) IV on day 1 of weeks 1, 5, and 9 (if mechlorethamine is unavailable, may substitute with cyclophosphamide [375 mg/m²] IV); etoposide (60 mg/m²) IV on days 1 and 2 of weeks 3, 7, and 11; and oral prednisone (40 mg/m²) every other day of weeks 1-9 followed by a taper. All patients with bulky disease receive radiotherapy 2-3 weeks after completion of chemotherapy.
Arm/Group | Arm A (ABVD) | Arm B (Stanford V)
Serious Adverse Events (participants affected / at risk) | 355/414 | 401/422
Other Adverse Events (participants affected / at risk) | 413/414 | 422/422
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (ABVD) (N=414) | Arm B (Stanford V) (N=422)
Allergic reaction (Immune system disorders) | 0 | 3
Allergy-other (Immune system disorders) | 0 | 1
Middle ear/hearing (Ear and labyrinth disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 20 | 86
Leukocytes decreased (Investigations) | 138 | 230
Lymphopenia (Investigations) | 175 | 328
Neutrophils decreased (Investigations) | 313 | 293
Platelets decreased (Investigations) | 10 | 9
Transfusion: pRBCs (Blood and lymphatic system disorders) | 3 | 16
Conduction abnormality (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 3
Supraventricular arrhythmias (Cardiac disorders) | 0 | 2
Cardiac-ischemia (Cardiac disorders) | 3 | 2
Cardiac-left ventricular function (Cardiac disorders) | 2 | 2
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 2
Pericardial effusion/pericarditis (Cardiac disorders) | 0 | 1
Peripheral arterial ischemia (Vascular disorders) | 0 | 2
Thrombosis/embolism (Vascular disorders) | 11 | 12
Cardiac-other (Cardiac disorders) | 1 | 1
Fatigue (General disorders) | 18 | 15
Fever (General disorders) | 7 | 8
Weight gain (Investigations) | 1 | 2
Coagulation-other (Investigations) | 0 | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1 | 1
Injection site reaction (General disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Radiation dermatitis (Injury, poisoning and procedural complications) | 0 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 3 | 1
Endocrine-other (Endocrine disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 13 | 15
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 5
Dysphagia-esophageal radiation (Gastrointestinal disorders) | 0 | 4
Gastritis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Mucositis due to radiation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 22 | 17
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 7
Vomiting (Gastrointestinal disorders) | 16 | 17
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 6
Hematemesis (Gastrointestinal disorders) | 0 | 1
Melena/GI bleeding (Gastrointestinal disorders) | 0 | 1
Alkaline phosphatase increased (Investigations) | 4 | 5
Blood bilirubin increased (Investigations) | 9 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 7
Aspartate aminotransferase increased (Investigations) | 4 | 4
Alanine aminotransferase increased (Investigations) | 0 | 1
Catheter-related infection (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 11
Infection w/ grade 3 or 4 neutropenia (Infections and infestations) | 23 | 27
Infection w/ unknown ANC (Infections and infestations) | 1 | 5
Infection w/o neutropenia (Infections and infestations) | 13 | 11
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 16
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Ataxia (Nervous system disorders) | 1 | 1
Delusions (Psychiatric disorders) | 0 | 1
Dizziness/lightheadedness (Nervous system disorders) | 1 | 1
Extrapyramidal movement (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 5
Anxiety/agitation (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 0 | 1
Neuropathy-cranial (Nervous system disorders) | 1 | 0
Neuropathy-motor (Nervous system disorders) | 3 | 24
Neuropathy-sensory (Nervous system disorders) | 11 | 39
Syncope (Nervous system disorders) | 4 | 5
Vertigo (Nervous system disorders) | 1 | 1
Blurred vision (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 11
Chest pain (General disorders) | 3 | 3
Dysmenorrhea (General disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Neuropathic pain (Nervous system disorders) | 3 | 5
Pain due to radiation (General disorders) | 0 | 1
Pain-other (General disorders) | 2 | 4
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
(DLCO) decreased (Investigations) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 14
FEV1 decreased (Investigations) | 0 | 2
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Voice changes/stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Creatinine increased (Investigations) | 5 | 9
Incontinence (Renal and urinary disorders) | 1 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1
Renal/GU-other (Renal and urinary disorders) | 1 | 0
Irregular menses (Reproductive system and breast disorders) | 1 | 11
Male infertility (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (ABVD) (N=414) | Arm B (Stanford V) (N=422)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 24 | 9
Anemia (Blood and lymphatic system disorders) | 374 | 412
Leukocytes decreased (Investigations) | 378 | 394
Lymphopenia (Investigations) | 319 | 379
Neutrophils decreased (Investigations) | 341 | 354
Platelets decreased (Investigations) | 118 | 116
Edema (Cardiac disorders) | 29 | 29
Phlebitis (Vascular disorders) | 25 | 35
Fatigue (General disorders) | 320 | 311
Fever (General disorders) | 62 | 57
Rigors/chills (General disorders) | 28 | 39
Sweating (Skin and subcutaneous tissue disorders) | 41 | 42
Weight gain (Investigations) | 34 | 47
Weight loss (Investigations) | 21 | 25
Alopecia (Skin and subcutaneous tissue disorders) | 287 | 318
Injection site reaction (General disorders) | 52 | 37
Nail changes (Skin and subcutaneous tissue disorders) | 31 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 31
Radiation dermatitis (Injury, poisoning and procedural complications) | 18 | 44
Rash/desquamation (Skin and subcutaneous tissue disorders) | 46 | 53
Hot flashes (Vascular disorders) | 30 | 24
Anorexia (Metabolism and nutrition disorders) | 83 | 66
Constipation (Gastrointestinal disorders) | 195 | 221
Dyspepsia (Gastrointestinal disorders) | 68 | 86
Dysphagia (Gastrointestinal disorders) | 48 | 82
Dysphagia-esophageal radiation (Gastrointestinal disorders) | 15 | 32
Mouth dryness (Gastrointestinal disorders) | 8 | 22
Nausea (Gastrointestinal disorders) | 313 | 283
Stomatitis (Gastrointestinal disorders) | 138 | 145
Taste disturbance (Nervous system disorders) | 54 | 47
Vomiting (Gastrointestinal disorders) | 191 | 135
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 75 | 56
Alkaline phosphatase increased (Investigations) | 156 | 108
Blood bilirubin increased (Investigations) | 25 | 35
Hypoalbuminemia (Metabolism and nutrition disorders) | 187 | 194
Aspartate aminotransferase increased (Investigations) | 115 | 111
Infection w/o neutropenia (Infections and infestations) | 83 | 57
Hyperglycemia (Metabolism and nutrition disorders) | 192 | 255
Hypoglycemia (Metabolism and nutrition disorders) | 51 | 35
Muscle weakness (Musculoskeletal and connective tissue disorders) | 10 | 22
Dizziness/lightheadedness (Nervous system disorders) | 32 | 39
Insomnia (Psychiatric disorders) | 67 | 140
Anxiety/agitation (Psychiatric disorders) | 32 | 46
Depression (Psychiatric disorders) | 34 | 23
Neuropathy-motor (Nervous system disorders) | 33 | 65
Neuropathy-sensory (Nervous system disorders) | 196 | 329
Abdominal pain (Gastrointestinal disorders) | 50 | 63
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 69
Bone pain (Musculoskeletal and connective tissue disorders) | 78 | 50
Chest pain (General disorders) | 34 | 35
Headache (Nervous system disorders) | 72 | 79
Myalgia (Musculoskeletal and connective tissue disorders) | 134 | 168
Pain-other (General disorders) | 32 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 117 | 59
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 110 | 95
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 30 | 15
Creatinine increased (Investigations) | 26 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No